CLINICAL TRIAL: NCT05001139
Title: A Multicenter, Open Label, Uncontrolled Study for the Evaluation of Efficacy and Safety by Clinical Parameters of Relizema Ecofoam in Adult Atopic and Contact Dermatitis
Brief Title: Clinical Investigation on the Efficacy and Safety of Relizema Ecofoam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Relife S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ReGl/20/Rec-Der/001
Record Dates: First submitted 2021-08-04; First posted 2021-08-11 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Dermatitis
Keywords: ecofoam
MeSH Terms: conditions — Dermatitis

STUDY DESIGN:
Intervention Model Description: Multicenter, open label, uncontrolled, single arm, post-market clinical folow-up study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relizema ecofoam (Experimental): Reizema ecofoam for 42 days, 2 times per day
  Interventions: Device: Relizema ecofoam

INTERVENTIONS:
Device: Relizema ecofoam — DermoRelizema ecofoam, class II a medical device, topical compact mousse, to be applied 2 times per day during the 42 days of study duration

SUMMARY:
The scope of this open label clinical trial is to evaluate and confirm the performance of Relizema ecofoam in the improvement of the dermatitis severity. The disease severity will be clinically measured through the Investigator Global Assessment (IGA) after 28 days of treatment.

DETAILED DESCRIPTION:
The scope of this open label clinical trial is to evaluate and confirm the performance of Relizema ecofoam in the improvement of the dermatitis severity, by alleviating the symptomatology. The product will be applied for 42 days of treatment, 2 times per day into the face.

The dermatologist will perform 3 clinical follow up visits to assess the efficacy and safety of the product

ELIGIBILITY:
Inclusion Criteria:

1. Subject's written informed consent obtained prior to any study-related procedures;
2. Generally healthy male and female aged ≥ 18 years;
3. Presence of atopic dermatitis (AD), irritant contact dermatitis (ICD) or allergic contact dermatitis (ACD) of mild-moderateseverity: ▪ IGA score 2 (=mild) or 3 (=moderate);
4. Dermatitis affecting one or more body areas (face, legs, arms, etc.);
5. Subjects with cooperative attitude, able to comprehend the full nature and the purpose of the investigation, including possible risks and side effects, and able to comply with the requirements of the entire investigation (including ability to attend the planned visits according to the time limits), based on Investigator's judgement.

Exclusion Criteria:

1. Severe dermatitis at inclusion;
2. Pregnant and breastfeeding women;
3. Concomitant other skin disorders including skin infections;
4. Currently or previously diagnosed or treated (chemotherapy and/or radiotherapy) for cancer in the past 5 years;
5. History of previous skin cancer (history of non-metastatic squamous or basal cell carcinoma of the skin is allowed);
6. Active infections or use of antibiotics in the past 7 days;
7. Diabetic subjects;
8. History of congenital or acquired immunodepression;
9. Immunologic or infectious disease (e.g. hepatitis, tuberculosis, HIV or AIDS, any typology of lupus, rheumatoid arthritis) which could place the subject at risk or interfere with study results;
10. Use of any topic medication for dermatitis in the past 14 days;
11. Use of any topic product for dermatitis in the 2 days before study treatment start;
12. Any systemic treatment or procedure that could influence dermatitis activity within the past 30 days (or 5 half-lives);
13. Use of any corticosteroids, immunosuppressant drugs or immunotherapy within the past 30 days (or 5 half-lives);
14. Use of oral antihistamines and antidepressants in the past 30 days;
15. Subjects with any other clinically significant or unstable concurrent disease or skin condition or general condition that, in the Investigator's opinion, might interfere with the study evaluations;
16. Allergy, sensitivity or intolerance to the components of the investigational device formulations ingredients;
17. Concomitant or previous participation in other interventional clinical study in the past 3 months;
18. Subjects planning sun exposure or tanning booths or UV sources throughout the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Micali, Principal Investigator — AOU Policlinico "G. Rodolico-San Marco" Catania
Locations (1):
- AOU Policlinico "G. Rodolico- San Marco", Catania, Italia, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Relizema Ecofoam
Started | 13
Completed | 7
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Relizema Ecofoam
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 13
Subjects affected by mild-to-moderate atopic and contact (irritant or allergic) dermatitis [Count of Participants; unit: Participants] | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Responded to Treatment With IGA Scale
Description: The disease severity will be clinically measured through the Investigator Global Assessment (IGA is based on a five-point scale:
  0 = clear
  1. = almost clear
  2. = mild 3= moderate
  4 = severe) for dermatitis after 28 days of treatment.
Time Frame: after 28 days of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Relizema Ecofoam
Number analyzed (Participants) | 7
Participants | 3

2. Secondary Outcome: Number of Participants Who Responded to Tretment
Description: to evaluate the performance of the Relizema ecofoam in the change of dermatitis severity (IGAs based on a five-point scale: 0 = clear
  1. = almost clear
  2. = mild 3= moderate
  4 = severe) after 42 days of treatment;
Time Frame: after 42 days of treatment
Population: Proportion of responders at visit 2 and visit 4, compared to baseline ( visit 1), visit 4 reported
Measure: Count of Participants; unit: Participants
Arm/Group | Relizema Ecofoam
Number analyzed (Participants) | 7
Participants | 3

3. Secondary Outcome: Eczema Area and Severity Index Code After 14, 28 and 42 Days of Treatment
Description: to evaluate the eczema change through the EASI (Eczema Area and Severity Index Four body regions are considered: head and neck, trunk (including genital area), upper limbs, lower limbs (including buttocks). The percentage of skin affected by eczema in each region is correlated to an area score (0 = 0: no eczema in this region, best result; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100%: the entire region is affected by eczema, worst result).
Time Frame: after 14, 28 and 42 days of treatment
Population: to evaluate the eczema change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relizema Ecofoam
Number analyzed (Participants) | 7
score on a scale
  after 14 days of treatment | 4.36 (4.83)
  after 28 days of treatment | 2.21 (2.34)
  after 42 days of treatment | 1.83 (1.20)

4. Secondary Outcome: Visual Analogue Scale Scores for Itching, Burning, Pain and Pruritus After 14, 28 and 42 Days of Treatment
Description: to evaluate the change in pain and pruritus at visits, as reported by the subject at visits by VAS (Visual Analogue Scale) The subject will be requested to indicate at each visit his/her itching, burning and pain by placing a vertical mark along a 100 mm VAS (Visual Analogue Scale).
  (0: best result, 100mm:worst result)
Time Frame: after 14, 28 and 42 days of treatment
Population: VAS for pain, burning and itching rating
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Relizema Ecofoam
Number analyzed (Participants) | 7
scores on a scale
  VAS for pain rating at Visit 1 | 13.42 (18.59)
  VAS for pian after 14 days of tratment | 15.33 (27.90)
  VAS for pian after 28 days of treatment | 8.71 (18.25)
  VAS for pain after 42 days of treatment | 20.83 (31.45)
  VAS for burning rating ai Visit 1 | 36.83 (36.80)
  VAS for burning after 14 days of treatment | 35 (37.67)
  VAS for burning after 28 days of treatment | 10.57 (18.12)
  VAS for burning after 42 days of treatment | 27.71 (30.72)
  VAS for itching ai visit 1 | 71.50 (26.89)
  VAS for itching after 14 days of treatment | 58.58 (40.27)
  VAS for itching after 28 days of treatment | 37.43 (32.91)
  VAS for itching after 42 days of treament | 52.17 (27.06)

5. Secondary Outcome: Quality of Life (QoL) Scores, After 14, 28 and 42 Days of Treatment
Description: to evaluate change in the Quality of Life (QoL) of the subject related to his/her dermatitis, through the DLQI (Dermatology Life Quality Index DLQI is a questionnaire used to measure the impact of skin disease on the quality of life of an affected person. There are 10 questions, covering the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, treatment. Each question refers to the impact of the skin disease on the patient's life over the previous week.
  Each question is scored from 0 to 3, giving a possible score range from 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).
  Global score:
  0-1 = No effect on patient's life 2-5 = Small effect 6-10 = Moderate effect 11-20 = Very large effect 21-30 = Extremely large effect. The DQLI will be compiled by the subject at each visit.) questionnaire;
Time Frame: after 14, 28 and 42 days of treatment
Population: DLQI score change from baseline (V1) to V2, V3 and V4.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Relizema Ecofoam
Number analyzed (Participants) | 7
scores on a scale
  At visit 1 | 5.08 (3.58)
  After 14 days of treatment | 4.33 (3.25)
  After 28 days of treatment | 2.52 (3.05)
  After 42 days of treatment | 3.50 (2.26)

6. Secondary Outcome: Unit on a Scale
Description: to evaluate the subject's adherence to treatment, reported on the subject's diary and the product accountability (100% is the best result, 0% is the worst)
Time Frame: after 14, 28 and 42 days of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Relizema Ecofoam
Number analyzed (Participants) | 7
units on a scale
  between visit 1 and visit 2 | 91.38 (17.10)
  between visit 2 and visit 3 | 97.14 (6.57)
  between visit 3 and visit 4 | 90.67 (15.52)

7. Secondary Outcome: to Evaluate the Subject's and Investigator's Global Evaluation of Performance of Relizema Ecofoam
Description: to evaluate the subject's and Investigator's global evaluation of performance of Relizema ecofoam by means of a 7-items scale (where 1 = very much improved, 2 = improved, 3 = minimally improved, 4
  = no change, 5 = minimally worse, 6 = worse, 7 = very much worse)
Time Frame: at the end of the study ( day 42)
Population: Subject's and Investigator's global evaluation on performance of the study product
Measure: Count of Participants; unit: Participants
Arm/Group | Relizema Ecofoam
Number analyzed (Participants) | 10
Participants
  improved or minimally improved | 3
  no changes | 1
  minimally worse, worse or very much worse | 6

8. Secondary Outcome: to Evaluate the Subject's Overall Acceptability of the Treatment
Description: to evaluate the subject's overall acceptability of the treatment (which takes into account pleasant or unpleasant feeling with the product and the ease of use), performed by means of a 5-item scale (where 1 = very much satisfied, 2 = satisfied, 3 = neither satisfied nor dissatisfied, 4 = dissatisfied, 5 = very much dissatisfied)
Time Frame: at the end of the study ( day 42)]
Population: Subject's evaluation of overall acceptability with treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Relizema Ecofoam
Number analyzed (Participants) | 10
Participants
  satisfied | 6
  neither satisfied neither dissatisfied | 1
  dissatisfied | 3

ADVERSE EVENTS:
Time Frame: 42 days
Arm/Group | Relizema Ecofoam
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT05001139/Prot_SAP_000.pdf